CLINICAL TRIAL: NCT06955117
Title: Comparative Study of McKenzie Technique and Manual Therapy for Pain and Function in Low Back Pain
Brief Title: McKenzie vs Manual Therapy for Low Back Pain
Acronym: LowBackpain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC01010SANA HAYAT
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy; Methods; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: one receiving McKenzie Technique and the other receiving Manual Therapy. Both groups will receive interventions independently to compare outcomes on pain and function in low back pain patients.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Technique (Group A) (Experimental): Experimental - McKenzie Technique (Group A) Intervention Type: Physical Therapy Intervention Name: McKenzie Extension Exercises
  Description:
  This group will receive McKenzie-based physical therapy including postural correction, prone lying, prone on elbows, prone press-ups (3×10), soft tissue mobilization (5-10 mins), lumbar mobilization (PA glide, side-lying rotations), METs (pelvic tilts, hip flexor stretch), core exercises (bridge, dead bug), plus hot pack (15-20 mins) and TENS (10 mins) before and after therapy.
  Interventions: Other: Physical Therapy Exercises
- Active Comparator: Manual Therapy (Group B) (Active Comparator): Physical Therapy Intervention Name: Manual Therapy and Exercises
  Description:
  Participants will receive soft tissue mobilization, lumbar mobilization (PA glide, side-lying rotations), METs (pelvic tilts, hip flexor stretch), core exercises (bridge, dead bug), general stretching, hot pack (15-20 mins), and TENS (10 mins) before mobilization. No McKenzie techniques will be applied.
  Interventions: Other: Physical Therapy Exercises; Other: Group B

INTERVENTIONS:
Other: Physical Therapy Exercises — Experimental - McKenzie Technique (Group A) Intervention Type: Other: Physical Therapy Exercises
  Other Names:
  Intervention for low back pain
  Description:
  Soft Tissue Mobilization: Manual massage to release muscle tension (5-10 mins)
  Lumbar Mobilization Techniques:
  PA Mobilization (Posteroanterior glide) on the lumbar spine (Grade I-IV, 3-5 min per segment)
  Side-lying Rotational Mobilization (3 sets × 10 reps)
  Muscle Energy Techniques (METs):
  Pelvic Tilts (3 sets × 10 reps)
  Hip Flexor Stretch with Isometric Hold (3 sets × 10 sec per side)
  Core Stabilization Exercises:
  Bridge Exercise (3 sets × 10-15 reps)
  Dead Bug Exercise (3 sets × 10 reps per side)
  Modalities:
  Hot Pack (15-20 mins) for relaxation before therapy
  TENS (10 mins) for pain relief before mobilization
  Other Names: intervention for low backpain
Other: Group B — Manual Therapy (Group B)
  Description:
  Soft Tissue Mobilization: Manual massage to release muscle tension (5-10 mins)
  Lumbar Mobilization Techniques:
  PA Mobilization (Posteroanterior glide) on the lumbar spine (Grade I-IV, 3-5 min per segment)
  Side-lying Rotational Mobilization (3 sets × 10 reps)
  Muscle Energy Techniques (METs):
  Pelvic Tilts (3 sets × 10 reps)
  Hip Flexor Stretch with Isometric Hold (3 sets × 10 sec per side)
  Core Stabilization Exercises:
  Bridge Exercise (3 sets × 10-15 reps)
  Dead Bug Exercise (3 sets × 10 reps per side)
  Modalities:
  Hot Pack (15-20 mins) for relaxation before therapy
  TENS (10 mins) for pain relief before mobilization
  Other Names: Manual Therapy (Group B)
  Arms: Active Comparator: Manual Therapy (Group B)

SUMMARY:
A comparative study evaluating the effectiveness of the McKenzie technique versus manual therapy in patients with nonspecific low back pain. The study aims to assess which intervention is more effective in reducing pain and improving functional mobility.

DETAILED DESCRIPTION:
The study compares McKenzie Method, a directional preference-based approach involving repeated movements and posture correction, against Manual Therapy, which includes hands-on techniques such as mobilizations and manipulations. Patients with nonspecific low back pain will be randomly assigned to one of the two groups and treated over a defined period. Outcomes will be measured using pain and disability scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonspecific low back pain lasting more than 4 weeks
* Willing to participate and comply with the study protocol

Exclusion Criteria:

* History of lumbar spine surgery
* Presence of spinal fracture, tumor, or infection
* Pregnant women
* Severe osteoporosis or spinal deformity

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-04-17 (Estimated); Study Completion 2027-04-17 (Estimated)

PRIMARY OUTCOMES:
To assess the change in pain intensity | 6 Months
  Pain intensity will be measured using the Visual Analog Scale (VAS), a 10-centimeter scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse outcomes. Pain levels will be assessed from baseline to the end of the intervention period.

SECONDARY OUTCOMES:
Disability score | 6months
  Disability will be assessed using the Oswestry Disability Index (ODI), a 0-100 scale, to evaluate the degree of functional limitation in daily activities.

OTHER OUTCOMES:
lumbar range of motion | 6 months
  Range of motion will be evaluated using goniometric measurements to assess changes in lumbar flexion and extension.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nadeem Ahmad, MS, Principal Investigator — Riphah International University Malakand Campus
Locations (1):
- Riphah international University Malakand, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No